CLINICAL TRIAL: NCT03265405
Title: Efficacy and Safety of Two Glucocorticoid Regimens in the Treatment of Sarcoidosis: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Two Glucocorticoid Regimens in the Treatment of Sarcoidosis
Acronym: SARCORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2017/299
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Sarcoidosis
Keywords: pulmonary sarcoidosis; corticosteroids; glucocorticoids; relapse; interstitial lung disease; diffuse parenchymal lung disease; immunosuppression; mediastinal lymphadenopathy
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary; Recurrence; Lung Diseases, Interstitial | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose prednisolone (Active Comparator): An initial dose of 20 mg/day will be administered for 8 weeks, followed by 15 mg/day for 8 weeks, 10 mg/day for 4 weeks, and 5 mg/day for 4 weeks, after which the drug will be tapered over 2 weeks and discontinued.
  Interventions: Drug: Low dose prednisolone
- Medium dose prednisolone (Active Comparator): An initial dose of 40 mg/day will be administered for 4 weeks, followed by 30 mg/day for 4 weeks, 20 mg/day for 4 weeks, 15 mg/day for 4 weeks, 10 mg/day for 4 weeks, and 5 mg/day for 4 weeks, after which the drug will be tapered over 2 weeks and discontinued.
  Interventions: Drug: Medium dose prednisolone

INTERVENTIONS:
Drug: Low dose prednisolone — An initial dose of 20 mg/day will be administered for 8 weeks, followed by 15 mg/day for 8 weeks, 10 mg/day for 4 weeks, and 5 mg/day for 4 weeks, after which the drug will be tapered over 2 weeks and discontinued.
  Arms: Low dose prednisolone
Drug: Medium dose prednisolone — An initial dose of 40 mg/day will be administered for 4 weeks, followed by 30 mg/day for 4 weeks, 20 mg/day for 4 weeks, 15 mg/day for 4 weeks, 10 mg/day for 4 weeks, and 5 mg/day for 4 weeks, after which the drug will be tapered over 2 weeks and discontinued.
  Arms: Medium dose prednisolone

SUMMARY:
For pulmonary sarcoidosis, the initial dose recommended by the joint statement of the American Thoracic Society (ATS), European Respiratory Society (ERS), and The World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) is 20-40 mg per day.5 The exact dose and duration of treatment for sarcoidosis are unknown.4 We hypothesize that a higher dose of 40 mg per day as compared to a 20 mg/day dose of prednisone will be more effective in preventing post-treatment relapse by effective initial suppression of the granulomatous inflammation and reduction of the disease load. In this study, we compare the efficacy and safety of medium dose (40 mg/day prednisone) and low dose (20 mg/day prednisone) glucocorticoids in the treatment of acute sarcoidosis.

DETAILED DESCRIPTION:
Glucocorticoids are the cornerstone of treatment of sarcoidosis and are used as the first-line agents in patients requiring immunosuppressive therapy.4 The optimal dose and duration of glucocorticoids is an unresolved issue. For pulmonary sarcoidosis, the initial dose recommended by the joint statement of the ATS/ERS/WASOG is 20-40 mg per day.5 The duration of treatment recommended is at least one year. However, mild disease of recent onset may respond to a shorter duration of treatment. Further, as most of the toxic effects of glucocorticoids are cumulative, the dose and duration of steroids need to be kept to a minimum to balance the benefit and risks of treatment.

Two large studies performed about two decades ago used an initial dose of 30 mg and 20 mg respectively for treating acute sarcoidosis. While the British Thoracic Society employed steroid treatment (initial dose 30 mg/day) for one year, in the Finnish study, oral glucocorticoids (initial dose 20 mg/day) were administered for three months and were followed by inhaled budesonide.3,6 In a recent Delphi study of experts, 37% and 20% of the experts used an initial prednisone equivalent dose of 40 mg per day and 20 mg per day regardless of weight, respectively.7 About 23% used doses of 20 mg, 30 mg, or 40 mg per day depending on weight. However, consensus was reached that a dose higher than 40 mg per day is not required. Apart from the initial response to glucocorticoids in symptoms and lung function, the rate of relapse after cessation of treatment is an important outcome in the management of sarcoidosis.

The exact dose and duration of treatment for sarcoidosis are unknown.4 We hypothesize that a higher dose of 40 mg per day as compared to a 20 mg/day dose of prednisone will be more effective in preventing post-treatment relapse by effective initial suppression of the granulomatous inflammation and reduction of the disease load. In this study, we compare the efficacy and safety of medium dose (40 mg/day prednisone) and low dose (20 mg/day prednisone) glucocorticoids in the treatment of acute sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Computed tomography of the chest consistent with a diagnosis of sarcoidosis of the lung/mediastinal lymph nodes
2. Diagnosis of sarcoidosis made on cytological or histological samples
3. Having significant symptoms requiring immunosuppressive treatment and/or having reduced lung function (defined as forced vital capacity or forced expiratory volume in one second (FEV1) less than 80% predicted) or an extrathoracic manifestation of the disease requiring treatment with low-medium dose glucocorticoids
4. Onset of symptoms within two years of study entry

Exclusion Criteria:

1. Pregnant or lactating women
2. Subjects having any manifestation requiring high dose steroid treatment (this includes symptomatic neurosarcoidosis, life threatening cardiac sarcoidosis, vision threatening posterior uveitis or other forms of vision threatening ocular sarcoidosis)
3. Having absolute contraindication for prednisone in a dose of 40 mg/day (this includes untreated glaucoma, uncontrolled diabetes mellitus, untreated infections, untreated severe psychiatric disorders)
4. Unwilling to participate in the study
5. Having received glucocorticoids (prednisolone equivalent >15 mg/day) for more than three weeks in the preceding two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Relapse or treatment failure | 18 months
  The proportion of subjects with a relapse or treatment failure in the two study groups (initial dose 40 mg/day versus 20 mg/day of prednisone) at the end of 18 months

SECONDARY OUTCOMES:
Mean time to relapse/treatment failure | 18 months
  The difference between the mean time to relapse/treatment failure in the study groups
Response | 18 months
  The proportion of subjects with worsening, stabilization, improvement or resolution of the disease in the study groups at the end of 18 months
Lung function early | 6 months
  The difference in the mean change in forced vital capacity between the study groups at the end of 6 months
Cumulative dose of prednisolone | 18 months
  The difference in the mean cumulative dose of prednisolone between the study groups at the end of 18 months
Adverse effects | 18 months
  The adverse effects of treatment (acne, weight gain, hyperglycemia, hypertension, adrenal insufficiency, osteoporosis and any other adverse effects related to prednisolone) between the study groups at the end of 18 months
Change in the sarcoidosis-related quality-of-life assessed by the score on the Sarcoidosis Health Questionnaire at treatment completion | 6 months
  The Sarcoidosis Health Questionnaire is a health-related quality-of-life questionnaire for patients with sarcoidosis. Higher scores reflect better quality-of-life
Change in the sarcoidosis-related quality-of-life assessed by the score on the Sarcoidosis Health Questionnaire at completion of follow-up | 18 months
  The Sarcoidosis Health Questionnaire is a health-related quality-of-life questionnaire for patients with sarcoidosis. Higher scores reflect better quality-of-life
Change in fatigue severity assessed by the score on the Fatigue Assessment Scale at treatment completion | 6 months
  The Fatigue Assessment Scale is a validated instrument for assessing sarcoidosis-related fatigue. Higher scores reflect more severe fatigue
Change in fatigue severity assessed by the score on the Fatigue Assessment Scale at completion of follow-up | 18 months
  The Fatigue Assessment Scale is a validated instrument for assessing sarcoidosis-related fatigue. Higher scores reflect more severe fatigue
Lung function late | 18 months
  The difference in the mean change in forced vital capacity between the study groups at the end of18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

REFERENCES:
- [Derived] Dhooria S, Sehgal IS, Agarwal R, Muthu V, Prasad KT, Dogra P, Debi U, Garg M, Bal A, Gupta N, Aggarwal AN. High-dose (40 mg) versus low-dose (20 mg) prednisolone for treating sarcoidosis: a randomised trial (SARCORT trial). Eur Respir J. 2023 Sep 9;62(3):2300198. doi: 10.1183/13993003.00198-2023. Print 2023 Sep. PMID 37690784